CLINICAL TRIAL: NCT01378065
Title: Restorelle Direct Fix A&P for Female Pelvic Organ Prolapse: A Prospective Post Market Study
Brief Title: Restorelle Direct Fix Anterior and Posterior (A&P) for Female Pelvic Organ Prolapse: A Prospective Post Market Study
Acronym: (A&P)
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: US011
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: POP; pelvic organ prolapse; anterior prolapse; posterior prolapse; vaginal prolapse; vaginal floor reconstruction
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Restorelle Direct Fix A&P — Restorelle Direct Fix A&P is a permanently implantable synthetic mesh for reconstruction of the pelvic floor secondary to the prolapse or protrusion of the pelvic organs into or out of the vaginal canal.

SUMMARY:
This is a prospective, multi-center study designed to assess the palpability of the Restorelle Direct Fix A&P mesh after vaginal reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult female at least 18 years of age
* Willing and able to provide written informed consent
* Diagnosed with clinically significant pelvic organ prolapse of Stage 2 or higher as determined by Pelvic Organ Prolapse Quantification System (POP-Q) requiring surgical intervention in the anterior and/or posterior compartment
* Willing and able to complete all follow-up visits and procedures indicated in the protocol

Exclusion Criteria:

* Concurrent surgical treatment of pelvic organ prolapse using anything other than the Restorelle Direct Fix A&P
* Confirmed Stage 2 or higher prolapse as determined by POP-Q for a compartment that is not being repaired in the same procedure
* Previous pelvic organ prolapse repair using synthetic grafts
* Patients requiring a total hysterectomy (i.e. removal of the cervix) at the time of vaginal reconstruction
* Patients requiring a procedure for fecal incontinence (i.e.) anal sphincteroplasty) at the time of vaginal reconstruction
* Pregnant or a desire to become pregnant
* Previous radiation or other treatments for cancer in the pelvic area
* Immunosuppression and/or current systemic steroid user
* On any anticoagulation therapy at the time of implant or with bleeding diathesis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects satisfying criteria for inclusion in the study were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Jarnagin, MD, Principal Investigator — Center for Pelvic Health, Franklin, TN, United States
Locations (6):
- United States (6):
  - MedStar Health Research Institute at Baltimore, Baltimore, Maryland
  - Female Pelvic Medicine & Urogynecology Institute of MI, Grand Rapids, Michigan
  - Central Missouri Women's Healthcare, Marshall, Missouri
  - Center for Pelvic Health, Franklin, Tennessee
  - The Group for Women, Norfolk, Virginia
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Restorelle Direct Fix: Subjects with clinically significant pelvic organ prolapse of Stage 2 or higher with surgical intervention using Restorelle Direct Fix A & P in the anterior and/or posterior compartment.
Period: Overall Study
Arm/Group | Restorelle Direct Fix
Started | 30 (31 subjects were enrolled/consented. However, 1 subject was not implanted with a study device.)
6 Week | 30
3 Months | 30
6 Months | 30
12 Months | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 27.9 (5.6)
Weight [Mean (Standard Deviation); unit: pound] | 164.7 (36.8)
Height [Mean (Standard Deviation); unit: Inches] | 64.3 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Palpability of the Restorelle Direct Fix Anterior and Posterior (A&P)
Description: Measured via palpability scale with possible outcomes of none, mild, moderate, or severe.
Time Frame: Baseline
Population: All subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Anterior - inside hymenal ring: None | 30
  Anterior - inside hymenal ring: Mild | 0
  Anterior - inside hymenal ring: Moderate | 0
  Anterior - inside hymenal ring: Severe | 0
  Anterior - 4 cm from introitus at midline: None | 30
  Anterior - 4 cm from introitus at midline: Mild | 0
  Anterior - 4 cm from introitus at midline: Moderat | 0
  Anterior - 4 cm from introitus at midline: Severe | 0
  Anterior - apex: None | 30
  Anterior - apex: Mild | 0
  Anterior - apex: Moderate | 0
  Anterior - apex: Severe | 0
  Posterior - inside hymenal ring: None | 30
  Posterior - inside hymenal ring: Mild | 0
  Posterior - inside hymenal ring: Moderate | 0
  Posterior - inside hymenal ring: Severe | 0
  Posterior - 4 cm from introitus at midline: None | 29
  Posterior - 4 cm from introitus at midline: Mild | 1
  Posterior - 4 cm from introitus at midline: Modera | 0
  Posterior - 4 cm from introitus at midline:Severe | 0
  Posterior - apex: None | 29
  Posterior - apex: Mild | 1
  Posterior - apex: Moderate | 0
  Posterior - apex: Severe | 0

2. Secondary Outcome: Rates of de Novo Dyspareunia
Description: Percentage of de novo dyspareunia measured via validated Participant Sexual Function Questionnaire-12 (PISQ-12) questionnaire at 6 weeks. The specific PISQ-12 score was based upon Question 3.5, "Do you feel pain during sexual intercourse?" The subjects' response was counted as having de novo dyspareunia if the response was "sometimes" "usually" or "always."
Time Frame: 6 weeks
Population: The 12 sexually active subjects without dyspareunia at baseline.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 12
percentage of subjects | 8.3

3. Secondary Outcome: Rates of de Novo Dyspareunia
Description: Percentage of de novo dyspareunia measured via validated Participant Sexual Function Questionnaire-12 (PISQ-12) questionnaire at 3 months. The specific PISQ-12 score was based upon Question 3.5, "Do you feel pain during sexual intercourse?" The subjects' response was counted as having de novo dyspareunia if the response was "sometimes" "usually" or "always."
Time Frame: 3 months
Population: The 12 sexually active subjects without dyspareunia at baseline.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 12
percentage of subjects | 8.3

4. Secondary Outcome: Rates of de Novo Dyspareunia
Description: Percentage of de novo dyspareunia measured via validated Participant Sexual Function Questionnaire-12 (PISQ-12) questionnaire at six months. The specific PISQ-12 score was based upon Question 3.5, "Do you feel pain during sexual intercourse?" The subjects' response was counted as having de novo dyspareunia if the response was "sometimes" "usually" or "always."
Time Frame: 6 months
Population: The 12 sexually active subjects without dyspareunia at baseline.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 12
percentage of subjects | 0

5. Secondary Outcome: Rates of de Novo Dyspareunia
Description: Percentage of de novo dyspareunia measured via validated Participant Sexual Function Questionnaire-12 (PISQ-12) questionnaire at 12 months. The specific PISQ-12 score was based upon Question 3.5, "Do you feel pain during sexual intercourse?" The subjects' response was counted as having de novo dyspareunia if the response was "sometimes" "usually" or "always."
Time Frame: 12 months
Population: The 11 sexually active subjects without dyspareunia at baseline. At the 12 month follow-up visit, only 11 subjects were sexually active and thus only 11 subjects completed Question 3.5 on the PISQ-12 questionnaire. Therefore, the number of participants analyzed for this outcome was 11 at the 12 month follow-up visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 11
percentage of subjects | 9.1

6. Secondary Outcome: Percentage of Participants With Surgical Success Rates of the Anterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at 6 Weeks
Description: Surgical success rates of the anterior compartments after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at 6 weeks. Surgical success rate is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 6 weeks
Population: The 27 subjects who were treated with Restorelle Direct Fix in the anterior compartment.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 27
percentage of subjects | 100

7. Secondary Outcome: Percentage of Participants With Surgical Success Rates of the Anterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at 3 Months
Description: Percentage of participants with surgical success rates of the anterior compartments after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at 3 months. Surgical success rate is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 3 months
Population: The 27 subjects who were treated with Restorelle Direct Fix in the anterior compartment.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 27
percentage of subjects | 100

8. Secondary Outcome: Percentage of Participants With Surgical Success Rates of the Anterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at 6 Months
Description: Percentage of participants with surgical success rates of the anterior compartments after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at 6 months. Surgical success rate is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 6 months
Population: The 27 subjects who were treated with Restorelle Direct Fix in the anterior compartment.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 27
percentage of subjects | 96.3

9. Secondary Outcome: Percentage of Participants With Surgical Success Rates of the Anterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at 12 Months
Description: Percentage of participants with surgical success rates of the anterior compartments after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at 12 months. Surgical success rate is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 12 months
Population: The 27 subjects who were treated with Restorelle Direct Fix in the anterior compartment.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 27
percentage of subjects | 100

10. Primary Outcome: Palpability of the Restorelle Direct Fix A&P
Description: Measured via palpability scale with possible outcomes of none, mild, moderate, or severe.
Time Frame: 6 weeks
Population: All subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Anterior - inside hymenal ring: None | 29
  Anterior - inside hymenal ring: Mild | 1
  Anterior - inside hymenal ring: Moderate | 0
  Anterior - inside hymenal ring: Severe | 0
  Anterior - 4 cm from introitus at midline: None | 27
  Anterior - 4 cm from introitus at midline: Mild | 3
  Anterior - 4 cm from introitus at midline: Moderat | 0
  Anterior - 4 cm from introitus at midline: Severe | 0
  Anterior - apex: None | 26
  Anterior - apex: Mild | 4
  Anterior - apex: Moderate | 0
  Anterior - apex: Severe | 0
  Posterior - inside hymenal ring: None | 30
  Posterior - inside hymenal ring: Mild | 0
  Posterior - inside hymenal ring: Moderate | 0
  Posterior - inside hymenal ring: Severe | 0
  Posterior - 4 cm from introitus at midline: None | 27
  Posterior - 4 cm from introitus at midline: Mild | 2
  Posterior - 4 cm from introitus at midline: Modera | 1
  Posterior - 4 cm from introitus at midline:Severe | 0
  Posterior - apex: None | 27
  Posterior - apex: Mild | 2
  Posterior - apex: Moderate | 1
  Posterior - apex: Severe | 0

11. Primary Outcome: Palpability of the Restorelle Direct Fix A&P
Description: Measured via palpability scale with possible outcomes of none, mild, moderate, or severe.
Time Frame: 3 months
Population: All study subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Anterior - inside hymenal ring: None | 29
  Anterior - inside hymenal ring: Mild | 1
  Anterior - inside hymenal ring: Moderate | 0
  Anterior - inside hymenal ring: Severe | 0
  Anterior - 4 cm from introitus at midline: None | 26
  Anterior - 4 cm from introitus at midline: Mild | 4
  Anterior - 4 cm from introitus at midline: Moderat | 0
  Anterior - 4 cm from introitus at midline: Severe | 0
  Anterior - apex: None | 26
  Anterior - apex: Mild | 4
  Anterior - apex: Moderate | 0
  Anterior - apex: Severe | 0
  Posterior - inside hymenal ring: None | 28
  Posterior - inside hymenal ring: Mild | 2
  Posterior - inside hymenal ring: Moderate | 0
  Posterior - inside hymenal ring: Severe | 0
  Posterior - 4 cm from introitus at midline: None | 28
  Posterior - 4 cm from introitus at midline: Mild | 2
  Posterior - 4 cm from introitus at midline: Modera | 0
  Posterior - 4 cm from introitus at midline:Severe | 0
  Posterior - apex: None | 28
  Posterior - apex: Mild | 2
  Posterior - apex: Moderate | 0
  Posterior - apex: Severe | 0

12. Primary Outcome: Palpability of the Restorelle Direct Fix A&P
Description: Measured via palpability scale with possible outcomes of none, mild, moderate, or severe.
Time Frame: 6 months
Population: All subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Anterior - inside hymenal ring: None | 30
  Anterior - inside hymenal ring: Mild | 0
  Anterior - inside hymenal ring: Moderate | 0
  Anterior - inside hymenal ring: Severe | 0
  Anterior - 4 cm from introitus at midline: None | 25
  Anterior - 4 cm from introitus at midline: Mild | 4
  Anterior - 4 cm from introitus at midline: Moderat | 1
  Anterior - 4 cm from introitus at midline: Severe | 0
  Anterior - apex: None | 25
  Anterior - apex: Mild | 2
  Anterior - apex: Moderate | 3
  Anterior - apex: Severe | 0
  Posterior - inside hymenal ring: None | 28
  Posterior - inside hymenal ring: Mild | 1
  Posterior - inside hymenal ring: Moderate | 1
  Posterior - inside hymenal ring: Severe | 0
  Posterior - 4 cm from introitus at midline: None | 26
  Posterior - 4 cm from introitus at midline: Mild | 3
  Posterior - 4 cm from introitus at midline: Modera | 1
  Posterior - 4 cm from introitus at midline:Severe | 0
  Posterior - apex: None | 27
  Posterior - apex: Mild | 1
  Posterior - apex: Moderate | 2
  Posterior - apex: Severe | 0

13. Primary Outcome: Palpability of the Restorelle Direct Fix A&P
Description: Measured via palpability scale with possible outcomes of none, mild, moderate, or severe.
Time Frame: 12 months
Population: All subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Anterior - inside hymenal ring: None | 29
  Anterior - inside hymenal ring: Mild | 1
  Anterior - inside hymenal ring: Moderate | 0
  Anterior - inside hymenal ring: Severe | 0
  Anterior - 4 cm from introitus at midline: None | 26
  Anterior - 4 cm from introitus at midline: Mild | 3
  Anterior - 4 cm from introitus at midline: Moderat | 1
  Anterior - 4 cm from introitus at midline: Severe | 0
  Anterior - apex: None | 26
  Anterior - apex: Mild | 4
  Anterior - apex: Moderate | 0
  Anterior - apex: Severe | 0
  Posterior - inside hymenal ring: None | 29
  Posterior - inside hymenal ring: Mild | 1
  Posterior - inside hymenal ring: Moderate | 0
  Posterior - inside hymenal ring: Severe | 0
  Posterior - 4 cm from introitus at midline: None | 28
  Posterior - 4 cm from introitus at midline: Mild | 2
  Posterior - 4 cm from introitus at midline: Modera | 0
  Posterior - 4 cm from introitus at midline:Severe | 0
  Posterior - apex: None | 27
  Posterior - apex: Mild | 3
  Posterior - apex: Moderate | 0
  Posterior - apex: Severe | 0

14. Secondary Outcome: Percentage of Participants With Mesh Exposure/Extrusion After Vaginal Reconstruction Surgery at 12 Months.
Description: Percentage of participants with anterior and posterior compartment mesh exposure/extrusion after vaginal reconstruction with Restorelle Direct Fix at 12 months. Per the protocol, mesh extrusion is defined as "passage gradually out of a body structure or tissue." Mesh exposure is defined as " a condition of displaying, revealing, exhibiting or making accessible e.g. vaginal mesh visualized through separated vaginal epithelium."
Time Frame: 12 months
Population: All study subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
percentage of subjects
  Rate of mesh exposure | 3.3
  Rate of mesh extrusion | 0.0

15. Secondary Outcome: Percentage of Participants With Surgical Success of the Posterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at the 6 Week Visit
Description: Percentage of participants with surgical success of the posterior compartment after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at the 6 week visit. Surgical success is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 6 week
Population: The 6 subjects who were treated in the posterior compartment with Restorelle Direct Fix.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 6
percentage of subjects | 100

16. Secondary Outcome: Percentage of Participants With Surgical Success of the Posterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at the 3 Month Visit
Description: Percentage of participants with surgical success of the posterior compartment after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at the 3 month visit. Surgical success is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 3 month
Population: The six subjects who had posterior compartment vaginal reconstruction surgery.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 6
percentage of subjects | 100

17. Secondary Outcome: Percentage of Participants With Surgical Success of the Posterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at the 6 Month Visit
Description: Percentage of participants with surgical success of the posterior compartment after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at the 6 month visit Surgical success is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 6 month
Population: The 5 subjects who were treated in the posterior compartment with Restorelle Direct Fix and have POP-Q measurement recorded at the six month follow-up visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 5
percentage of subjects | 100

18. Secondary Outcome: Percentage of Participants With Surgical Success of the Posterior Compartment After Vaginal Reconstruction Surgery Via Pelvic Organ Prolapse Quantification System (POP-Q) at the12 Month Visit
Description: Percentage of participants with surgical success of the posterior compartment after vaginal reconstruction surgery via Pelvic Organ Prolapse Quantification system (POP-Q) at the 12 month visit. Surgical success is defined as the post-operative point of maximal prolapse being less than 0 cm (i.e. above the hymenal ring).
Time Frame: 12 month
Population: The 6 subjects who were treated in the posterior compartment with Restorelle Direct Fix.
Measure: Number; unit: percentage of subjects
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 6
percentage of subjects | 100

19. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Questionnaire Since Treatment at 6 Weeks.
Description: The PGI-I Index consists on one question and was collected at 6 weeks. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation." There are seven possible responses including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse" and the subject chooses one response.
Time Frame: 6 weeks
Population: The 29 subjects who completed the PGI-I at the six week follow up visit.
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 29
participants
  Very much better | 15
  Much better | 10
  A little better | 1
  No change | 1
  A little worse | 0
  Much worse | 2
  Very much worse | 0

20. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Index Since Treatment at 3 Months.
Description: The PGI-I Index consists on one question and was collected at 3 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation. There are seven possible responses including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse" and the subject chooses one response.
Time Frame: 3 months
Population: The 29 subjects who completed the PGI-I at the three month follow up visit.
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 29
participants
  Very much better | 14
  Much better | 9
  A little better | 2
  No change | 3
  A little worse | 1
  Much worse | 0
  Very much worse | 0

21. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Index Since Treatment at 6 Months.
Description: The PGI-I Index consists on one question and was collected at 6 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation. There are seven possible responses including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse" and the subject chooses one response.
Time Frame: 6 months
Population: The 29 subjects who completed the PGI-I at the six month follow up visit.
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 29
participants
  Very much better | 12
  Much better | 7
  A little better | 6
  No change | 2
  A little worse | 1
  Much worse | 1
  Very much worse | 0

22. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Index Since Treatment at 12 Months.
Description: The PGI-I Index consists on one question and was collected at 12 months. The question is "Check the box that best describes how your condition is now, compared with how it was before you had the operation. There are seven possible responses including "very much better," "much better," "a little better," "no change," "a little worse," "much worse" and "very much worse" and the subject chooses one response.
Time Frame: 12 months
Population: All subjects
Measure: Number; unit: participants
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
participants
  Very much better | 18
  Much better | 4
  A little better | 4
  No change | 3
  A little worse | 1
  Much worse | 0
  Very much worse | 0

23. Secondary Outcome: Bladder Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Urinary Distress Inventory-6 (UDI-6) Questionnaire at 6 Weeks
Description: Bladder function is measured by UDI-6 Questionnaire at 6 weeks. The UDI-6 measures bladder function. The range of responses is: 1-4 with (1) not at all, (2) somewhat, (3) moderately, and (4 quite a bit). To allow for missing responses, the average score of items responded to, rather than the total, is taken. The average, which ranges from 1 to 4, is multiplied by 25 to put scores on a scale of 0 to 100. Higher scores indicate worse symptoms.
Time Frame: Baseline and 6 weeks
Population: All subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 45.1 (27.2)
  6 weeks | 25.7 (19.0)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p < .001, t-test, 2 sided

24. Secondary Outcome: Bladder Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Urinary Distress Inventory-6 (UDI-6) Questionnaire at 3 Months
Description: Bladder function is measured by UDI-6 Questionnaire at 3 months. The UDI-6 measures bladder function. The range of responses is: 1-4 with (1) not at all, (2) somewhat, (3) moderately, and (4 quite a bit). To allow for missing responses, the average score of items responded to, rather than the total, is taken. The average, which ranges from 1 to 4, is multiplied by 25 to put scores on a scale of 0 to 100. Higher scores indicate worse symptoms.
Time Frame: Baseline and 3 months
Population: All subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 45.1 (27.2)
  3 months | 17.1 (17.3)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p < .001, t-test, 2 sided

25. Secondary Outcome: Bladder Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Urinary Distress Inventory-6 (UDI-6) Questionnaire at 6 Months
Description: Bladder function is measured by UDI-6 Questionnaire at 6 months. The UDI-6 measures bladder function. The range of responses is: 1-4 with (1) not at all, (2) somewhat, (3) moderately, and (4 quite a bit). To allow for missing responses, the average score of items responded to, rather than the total, is taken. The average, which ranges from 1 to 4, is multiplied by 25 to put scores on a scale of 0 to 100. Higher scores indicate worse symptoms.
Time Frame: Baseline and 6 months
Population: All subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 45.1 (27.2)
  6 months | 16.4 (18.7)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p < .001, t-test, 2 sided

26. Secondary Outcome: Bladder Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Urinary Distress Inventory-6 (UDI-6) Questionnaire at 12 Months
Description: Bladder function is measured by UDI-6 Questionnaire at 12 months. The UDI-6 measures bladder function. The range of responses is: 1-4 with (1) not at all, (2) somewhat, (3) moderately, and (4 quite a bit). To allow for missing responses, the average score of items responded to, rather than the total, is taken. The average, which ranges from 1 to 4, is multiplied by 25 to put scores on a scale of 0 to 100. Higher scores indicate worse symptoms.
Time Frame: Baseline and 12 months
Population: All subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 45.1 (27.2)
  12 months | 18.1 (21.3)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p < .001, t-test, 2 sided

27. Secondary Outcome: Sexual Function After Vaginal Reconstruction With Restorelle Direct Fix Measured by Participant Sexual Function Questionnaire-12 (PISQ-12) at 6 Weeks
Description: Sexual function in women with pelvic organ prolapse is measured by the PISQ-12 at 6 weeks. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Time Frame: Baseline and 6 weeks
Population: The 28 subjects who completed the PISQ-12 at the six week follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 28
units on a scale
  Baseline | 15.7 (6.2)
  6 weeks | 14.7 (4.9)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p = 0.202, t-test, 2 sided

28. Secondary Outcome: Sexual Function After Vaginal Reconstruction With Restorelle Direct Fix Measured by Participant Sexual Function Questionnaire-12 (PISQ-12) at 3 Months
Description: Sexual function in women with pelvic organ prolapse is measured by the PISQ-12 at 3 months. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Time Frame: Baseline and 3 months
Population: The 25 subjects who completed the PISQ-12 at the three month follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 25
units on a scale
  3 month | 12.2 (5.2)
  Baseline | 15.7 (6.2)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

29. Secondary Outcome: Sexual Function After Vaginal Reconstruction With Restorelle Direct Fix Measured by Participant Sexual Function Questionnaire-12 (PISQ-12) at 6 Months
Description: Sexual function in women with pelvic organ prolapse is measured by the PISQ-12 at 6 months. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Time Frame: Baseline and 6 months
Population: The 26 subjects who completed the PISQ-12 at the six month follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 26
units on a scale
  6 months | 12.8 (5.4)
  Baseline | 15.7 (6.2)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

30. Secondary Outcome: Sexual Function After Vaginal Reconstruction With Restorelle Direct Fix Measured by Participant Sexual Function Questionnaire-12 (PISQ-12) at 12 Months
Description: Sexual function in women with pelvic organ prolapse is measured by the PISQ-12 at12 months. The scores range from 0-48 with lower scores indicating better sexual function. Scores are calculated by totalling the scores for each question with (4) always, (3) usually, (2) sometimes, (1) seldom, and (0) never. Reverse scoring is used for items 1, 2, 3 and 4. The short form questionnaire can be used with up to two missing responses. To handle missing values, the sum is calculated by multiplying the number of items by the mean of the answered items.
Time Frame: Baseline and 12 months
Population: The 25 subjects who completed the PISQ-12 at the twelve month follow up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 25
units on a scale
  12 month | 12.8 (6.2)
  Baseline | 15.7 (6.2)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Test type: Superiority or Other; p = 0.034, t-test, 2 sided

31. Secondary Outcome: Bowel Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Colorectal-Anal Distress Inventory 8 (CRADI-8) Questionnaire at the 6 Week Visit
Description: Colorectal-anal Distress Inventory is measured by the CRADI-8 at 6 weeks. The range of responses is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress).
Time Frame: Baseline and 6 weeks
Population: All subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 24.9 (20.7)
  6 weeks | 15.7 (15.7)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Analysis baseline to 6 weeks; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

32. Secondary Outcome: Bowel Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Colorectal-Anal Distress Inventory 8 (CRADI-8) Questionnaire at the 3 Month Visit
Description: Colorectal-anal Distress Inventory is measured by the CRADI-8 at 3 months. The range of responses is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress).
Time Frame: Baseline and 3 months
Population: All subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 24.9 (20.7)
  3 months | 15.3 (16.7)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Analysis baseline to 3 months; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

33. Secondary Outcome: Bowel Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Colorectal-Anal Distress Inventory 8 (CRADI-8) Questionnaire at the 6 Month Visit
Description: Colorectal-anal Distress Inventory is measured by the CRADI-8 at 6 months. The range of responses is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress).
Time Frame: Baseline and 6 months
Population: All subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 24.9 (20.7)
  6 months | 14.1 (16.1)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Analysis baseline to 6 months; Test type: Superiority or Other; p < .001, t-test, 2 sided

34. Secondary Outcome: Bowel Function After Vaginal Reconstruction Surgery With Restorelle Direct Fix A & P Measured by Colorectal-Anal Distress Inventory 8 (CRADI-8) Questionnaire at the12 Month Visit
Description: Colorectal-anal Distress Inventory is measured by the CRADI-8 at 12 months. The range of responses is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Scores are calculated by multiplying the mean value of all questions answered by 25. The range of responses is: 0-100 with 0 (least distress) to 100 (most distress).
Time Frame: Baseline and 12 months
Population: All subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle Direct Fix
Number analyzed (Participants) | 30
units on a scale
  Baseline | 24.9 (20.7)
  12 months | 10.8 (14.0)
Statistical Analysis 1: Comparison: Restorelle Direct Fix; Analysis baseline to 12 months; Test type: Superiority or Other; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Restorelle Direct Fix
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restorelle Direct Fix (N=30)
Recurrent prolapse: Anterior Stage 2 (Reproductive system and breast disorders) | 1 (1) — Patient lifted heavy boxes during the post-operative period, but did not report this until her 12 month visit at which time she was referred for sacral colpopexy.
Right ureteral obstruction, hydronephrosis (Reproductive system and breast disorders) | 1 (1) — Hydronephrosis following gyn surgery. Right ureteral obstruction, secondary to suture holding distal arm behind pubic symphysis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restorelle Direct Fix (N=30)
Recurrent anterior prolapse (Reproductive system and breast disorders) | 2 (2) — One patient had Stage 1 and one patient had Stage 2 prolapse.
Wound dehiscence (Reproductive system and breast disorders) | 1 (1) — Subject had a small apical wound dehiscence with mesh exposure. The wound dehiscence was treated with a porcine graft.

LIMITATIONS AND CAVEATS:
The study N was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less